CLINICAL TRIAL: NCT04052321
Title: Quantification of Chest Wall Changes After Nuss Bar Removal Utilizing Three-dimensional Optical Surface Scans
Acronym: CHEST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: METCZ20190103
Record Dates: First submitted 2019-08-02; First posted 2019-08-09 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-07

CONDITIONS: Pectus Excavatum
Keywords: Three-dimensional optical surface imaging; Chest wall changes
MeSH Terms: conditions — Funnel Chest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3D scan arm (Experimental): This is a single arm study. Patients in this arm will receive a 3D scan just prior to, 2 weeks after, as well as 6 and 12 months after Nuss bar removal.
  Interventions: Other: 3D optical surface scan

INTERVENTIONS:
Other: 3D optical surface scan — A 3D optical surface scan is acquired utilizing a handheld 3D scanner. Such a scanner is comparable to an ordinary photo camera, however, it also records depth.

SUMMARY:
Pectus excavatum is the most common anterior chest wall deformity that affects up to 1:400 of newborns. If an operative correction is indicated, patients are often operated via the Ravitsch or Nuss bar procedure. The latter (i.e. the Nuss bar procedure) is the most commonly performed procedure. During this procedure one or more metal bars are inserted behind the sternum to push the sternum back into its normal position. These bars remain in situ for two-to-three years before being removed. Despite the fact that the Nuss bar procedure is regarded as an effective procedure, retraction may occur after removal. A recent study has investigated this phenomenon, utilizing three-dimensional (3D) optical surface scans acquired before and after Nuss bar removal. The authors found statistically significant changes to occur in chest wall dimensions directly after, as well as between 2 and 8 weeks after Nuss bar explantation, in comparison to the situation just prior to bar removal. They, moreover, found the time the bar was in situ to be predictive for retraction. However, the authors also stressed that further studies are needed to reinforce their preliminary findings and perform long-term assessments. Subsequently, a similar study with long-term assessments will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Patients that received 1 or more Nuss bar(s) to treat pectus excavatum and is/are scheduled to be removed due to the end of treatment.

Exclusion Criteria:

* Patients in which the Nuss bar(s) or its stabilizers are or have been dislocated.
* Patients that received a second operation to treat any complications regarding the initial Nuss bar implantation.
* Patients with proven connective tissue diseases (e.g. Marfan's syndrome).
* Patients with a diagnosis of epilepsy (as the 3D scanner utilizes flashing light to acquire the torso topography)
* Patients that are not fit to remain in a standing position with their arms above shoulder level for a maximum of 60 seconds.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Mean change in distance | Changes from baseline (prior to surgery) to the situation 2 weeks after surgery, as well as after 6 and 12 months
  The mean distance of thoracic wall changes
Maximum change in distance | Changes from baseline (prior to surgery) to the situation 2 weeks after surgery, as well as after 6 and 12 months
  The maximum distance of thoracic wall changes
Volumetric changes | Changes from baseline (prior to surgery) to the situation 2 weeks after surgery, as well as after 6 and 12 months
  The volumetric chest wall changes

SECONDARY OUTCOMES:
Predictors of chest wall changes | Changes in volume, mean and maximum distance from baseline to 12 months
  Predictors of chest wall changes, assessed by multivariate analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Zuyderland Medical Centre, Heerlen, Limburg, Netherlands

REFERENCES:
- [Background] Gomes-Fonseca J, Vilaca JL, Henriques-Coelho T, Direito-Santos B, Pinho ACM, Fonseca JC, Correia-Pinto J. A new methodology for assessment of pectus excavatum correction after bar removal in Nuss procedure: Preliminary study. J Pediatr Surg. 2017 Jul;52(7):1089-1097. doi: 10.1016/j.jpedsurg.2016.12.029. Epub 2017 Jan 7. PMID 28094014